CLINICAL TRIAL: NCT00761657
Title: A Randomized, Single-blind, Placebo-controlled, 4-Week Treatment Study of the Safety and Biologic Activity of Escalating Multiple Oral Doses of FG-4592 in Subjects With Chronic Kidney Disease Not Requiring Dialysis
Brief Title: Phase 2 Study of Roxadustat in Participants With Anemia and Chronic Kidney Disease Not Requiring Dialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FGCL-SM4592-017
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Results first posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Chronic Kidney Disease; Anemia
Keywords: Kidney; Chronic Kidney Disease; CKD; Stage 3 or 4 Chronic Kidney Disease; Renal; Anemia; Oral anemia treatment; Hemoglobin levels; Blood count; Erythropoietin
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — roxadustat

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Roxadustat 0.7 mg/kg BIW (Experimental): Participants will receive roxadustat 0.7 mg/kg BIW orally with doses administered at least 68 hours apart for 29 days.
  Interventions: Drug: Roxadustat
- Roxadustat 0.7 mg/kg TIW (Experimental): Participants will receive roxadustat 0.7 mg/kg TIW orally with doses administered at least 46 hours apart for 26 days.
  Interventions: Drug: Roxadustat
- Roxadustat 1.0 mg/kg BIW (Experimental): Participants will receive roxadustat 1.0 mg/kg BIW orally with doses administered at least 72 hours apart for 29 days.
  Interventions: Drug: Roxadustat
- Roxadustat 1.0 mg/kg TIW (Experimental): Participants will receive roxadustat 1.0 mg/kg TIW orally with doses administered at least 48 hours apart for 26 days.
  Interventions: Drug: Roxadustat
- Roxadustat 1.5 mg/kg BIW (Experimental): Participants will receive roxadustat 1.5 mg/kg BIW orally with doses administered at least 68 hours apart for 29 days.
  Interventions: Drug: Roxadustat
- Roxadustat 1.5 mg/kg TIW (Experimental): Participants will receive roxadustat 1.5 mg/kg TIW orally with doses administered at least 46 hours apart for 26 days.
  Interventions: Drug: Roxadustat
- Roxadustat 2.0 mg/kg BIW (Experimental): Participants will receive roxadustat 2.0 mg/kg BIW orally with doses administered at least 68 hours apart for 29 days.
  Interventions: Drug: Roxadustat
- Roxadustat 2.0 mg/kg TIW (Experimental): Participants will receive roxadustat 2.0 mg/kg TIW orally with doses administered at least 46 hours apart for 26 days.
  Interventions: Drug: Roxadustat
- Placebo (Placebo Comparator): Participants will receive placebo orally, matching to the roxadustat dose, number of days per week, and duration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roxadustat — Capsule
  Other Names: FG-4592
  Arms: Roxadustat 0.7 mg/kg BIW; Roxadustat 0.7 mg/kg TIW; Roxadustat 1.0 mg/kg BIW; Roxadustat 1.0 mg/kg TIW; Roxadustat 1.5 mg/kg BIW; Roxadustat 1.5 mg/kg TIW; Roxadustat 2.0 mg/kg BIW; Roxadustat 2.0 mg/kg TIW
Drug: Placebo — Capsule
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the safety, tolerability, and pharmacodynamic effects of different oral doses of roxadustat administered 2 times a week (BIW) or 3 times a week (TIW) for up to 4 weeks to participants with chronic kidney disease (CKD) not requiring dialysis.

DETAILED DESCRIPTION:
This study in participants with CKD not requiring dialysis was conducted in 2 parts (designated Part 1 and Part 2). Part 1 evaluated roxadustat doses at 1.0 and 2.0 milligrams/kilograms (mg/kg). Part 2 evaluated roxadustat doses at 0.7, 1.5, and 2.0 mg/kg.

On 08 May 2007, the Food and Drug Administration (FDA) placed a clinical hold on the study until evaluation of a report of a death due to fulminant hepatic failure in a participant with CKD in a FibroGen-sponsored clinical trial of another hypoxia inducible factor-prolyl hydroxylase inhibitor (HIF-PHI) (FG-2216) being investigated for treatment of anemia in participants with CKD and other diseases. The clinical hold resulted in early termination of Part 1 of the study. On 24 March 2008, the FDA lifted the clinical hold and Part 2 of this study started.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age. Participants aged over 75 years but otherwise meet all other participant selection criteria will be evaluated on a case-by-case basis and can be included in this study, per discretion of Sponsor's physician representative such as medical monitor or clinical leader.
2. Chronic Kidney Disease Stage 3 or 4 with hemoglobin <11.0 grams (g)/deciliter (dL).
3. Normal iron studies.
4. Normal folate and vitamin B12 levels.
5. Liver function tests within normal limits at screening.
6. Absence of active or chronic rectal bleeding.
7. Absence of diagnosis of age-related macular degeneration (AMD), diabetic macular edema, or diabetic proliferative retinopathy that is likely to require treatment during the trial.
8. Female participants must not be pregnant nor breastfeeding and agree to use acceptable method of contraception.
9. Male participants with partners who can have children must agree to use a medically acceptable method of contraception.

Exclusion Criteria:

1. Seropositive for HIV.
2. History of chronic liver disease.
3. History of polycystic kidney disease (PKD).
4. Uncontrolled hypertension (diastolic BP >110 millimeter of mercury (mmHg) or systolic BP >170 mmHg at screening).
5. New York Heart Association Class III or IV congestive heart failure.
6. Recent myocardial infarction or acute coronary syndrome.
7. History of myelodysplastic syndrome.
8. Any history of malignancy or a known genetic predisposition for developing cancer (for example, with diagnostic markers suggesting a genetic predisposition of cancer) except for curatively resected basal cell carcinoma of skin, squamous cell carcinoma of skin, cervical carcinoma in situ, or resected benign colonic polyps.
9. Active inflammatory infection or chronic inflammatory disease.
10. Any clinically significant and uncontrolled medical condition considered a high risk for participation in an investigational study.
11. Blood clots within 4 weeks.
12. History of ongoing hemolysis or diagnosis of hemolytic syndrome.
13. Known history of bone marrow fibrosis.
14. History of hemosiderosis or hemochromatosis.
15. Androgen therapy within 12 weeks.
16. Red blood cell transfusion within 12 weeks.
17. Therapy with an erythropoiesis stimulating agent (ESA) such as human recombinant erythropoietin within the past 60 days.
18. Intravenous iron supplementation within the past 60 days.
19. Currently taking dapsone or acetaminophen >2.6 g/day.
20. History of prior organ transplantation.
21. Alcohol consumption greater than 3 or more drinks per day within the past year.
22. Use of an investigational medication or participation in an investigational study within 4 weeks preceding Day 1.
23. Positive urine toxicology screen for a substance that has not been prescribed for the participant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2006-11-01 (Actual); Primary Completion 2010-06-21 (Actual); Study Completion 2010-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Peoria, Arizona
  - Tempe, Arizona
  - Los Angeles, California
  - Mission Viejo, California
  - Sacramento, California
  - San Diego, California
  - Whittier, California
  - Arvada, Colorado
  - Westminster, Colorado
  - Middlebury, Connecticut
  - Ocala, Florida
  - Panama City, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - Evergreen Park, Illinois
  - Wichita, Kansas
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Shreveport, Louisiana
  - Detroit, Michigan
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Flushing, New York
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Toledo, Ohio
  - Medford, Oregon
  - Wynnewood, Pennsylvania
  - Columbia, South Carolina
  - Orangeburg, South Carolina
  - Chattanooga, Tennessee
  - Houston, Texas

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Besarab A, Provenzano R, Hertel J, Zabaneh R, Klaus SJ, Lee T, Leong R, Hemmerich S, Yu KH, Neff TB. Randomized placebo-controlled dose-ranging and pharmacodynamics study of roxadustat (FG-4592) to treat anemia in nondialysis-dependent chronic kidney disease (NDD-CKD) patients. Nephrol Dial Transplant. 2015 Oct;30(10):1665-73. doi: 10.1093/ndt/gfv302. Epub 2015 Aug 3. PMID 26238121

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: On 08 May 2007, the Food and Drug Administration (FDA) placed a clinical hold on the study. The clinical hold resulted in early termination of Part 1 of the study. On 24 March 2008, the FDA lifted the clinical hold and Part 2 of this study started.
Groups:
- Roxadustat 0.7 Milligrams/Kilograms (mg/kg) BIW: Participants received roxadustat 0.7 mg/kg BIW orally with doses administered at least 68 hours apart for 29 days.
- Roxadustat 0.7 mg/kg TIW: Participants received roxadustat 0.7 mg/kg TIW orally with doses administered at least 46 hours apart for 26 days.
- Roxadustat 1.0 mg/kg BIW: Participants received roxadustat 1.0 mg/kg BIW orally with doses administered at least 72 hours apart for 29 days.
- Roxadustat 1.0 mg/kg TIW: Participants received roxadustat 1.0 mg/kg TIW orally with doses administered at least 48 hours apart for 26 days.
- Roxadustat 1.5 mg/kg BIW: Participants received roxadustat 1.5 mg/kg BIW orally with doses administered at least 68 hours apart for 29 days.
- Roxadustat 1.5 mg/kg TIW: Participants received roxadustat 1.5 mg/kg TIW orally with doses administered at least 46 hours apart for 26 days.
- Roxadustat 2.0 mg/kg BIW: Participants received roxadustat 2.0 mg/kg BIW orally with doses administered at least 68 hours apart for 29 days.
- Roxadustat 2.0 mg/kg TIW: Participants received roxadustat 2.0 mg/kg TIW orally with doses administered at least 46 hours apart for 26 days.
- Placebo: Participants received placebo orally, matching to the roxadustat dose, number of days per week, and duration.
Period: Part 1 (up to Day 57)
Arm/Group | Roxadustat 0.7 Milligrams/Kilograms (mg/kg) BIW | Roxadustat 0.7 mg/kg TIW | Roxadustat 1.0 mg/kg BIW | Roxadustat 1.0 mg/kg TIW | Roxadustat 1.5 mg/kg BIW | Roxadustat 1.5 mg/kg TIW | Roxadustat 2.0 mg/kg BIW | Roxadustat 2.0 mg/kg TIW | Placebo
Started | 0 | 0 | 12 | 10 | 0 | 0 | 1 | 2 | 10
Safety Population (Participants who received at least 1 dose of study drug.) | 0 | 0 | 12 | 9 | 0 | 0 | 1 | 2 | 10
Efficacy Evaluable (EE) Population (Participants who were anemic at baseline (hemoglobin [Hb] ≤11.0 grams/deciliter (g/dL) and were in study treatment for at least 2.5 weeks with corresponding Hb values.) | 0 | 0 | 5 | 5 | 0 | 0 | 0 | 1 | 6
Pharmacokinetic (PK) Population (Participants treated with roxadustat at the 2 PK sites.) | 0 | 0 | 5 | 3 | 0 | 0 | 1 | 2 | 0
Completed | 0 | 0 | 8 | 4 | 0 | 0 | 0 | 1 | 9
Not Completed | 0 | 0 | 4 | 6 | 0 | 0 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 3 | 4 | 0 | 0 | 1 | 1 | 1
Period: Part 2 (up to Day 114)
Arm/Group | Roxadustat 0.7 Milligrams/Kilograms (mg/kg) BIW | Roxadustat 0.7 mg/kg TIW | Roxadustat 1.0 mg/kg BIW | Roxadustat 1.0 mg/kg TIW | Roxadustat 1.5 mg/kg BIW | Roxadustat 1.5 mg/kg TIW | Roxadustat 2.0 mg/kg BIW | Roxadustat 2.0 mg/kg TIW | Placebo
Started | 10 | 13 | 0 | 0 | 10 | 11 | 10 | 10 | 18
Safety Population (Participants who received at least 1 dose of study drug.) | 10 | 13 | 0 | 0 | 10 | 11 | 10 | 10 | 18
EE Population (Participants who were anemic at baseline (hemoglobin [Hb] ≤11.0 grams/deciliter (g/dL) and were in study treatment for at least 2.5 weeks with corresponding Hb values.) | 10 | 12 | 0 | 0 | 10 | 11 | 10 | 10 | 11
PK Population (Participants who received roxadustat and had sufficient plasma data to allow calculation of PK parameters.) | 10 | 13 | 0 | 0 | 10 | 11 | 10 | 10 | 0
Completed | 10 | 13 | 0 | 0 | 10 | 11 | 10 | 10 | 17
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Part 1 and Part 2 Safety Population: Participants who received at least 1 dose of study drug.
Groups:
- Roxadustat 0.7 mg/kg BIW: Participants received roxadustat 0.7 mg/kg BIW orally with doses administered at least 68 hours apart for 29 days.
- Total: Total of all reporting groups
Arm/Group | Roxadustat 0.7 mg/kg BIW | Roxadustat 0.7 mg/kg TIW | Roxadustat 1.0 mg/kg BIW | Roxadustat 1.0 mg/kg TIW | Roxadustat 1.5 mg/kg BIW | Roxadustat 1.5 mg/kg TIW | Roxadustat 2.0 mg/kg BIW | Roxadustat 2.0 mg/kg TIW | Placebo | Total
Number analyzed (Participants) | 10 | 13 | 12 | 9 | 10 | 11 | 11 | 12 | 28 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (4.9) | 60.6 (9.2) | 69.5 (7.7) | 67.0 (8.4) | 63.8 (8.8) | 63.5 (6.4) | 64.3 (9.0) | 66.8 (7.8) | 68.6 (6.2) | 65.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 8 | 3 | 6 | 10 | 8 | 9 | 12 | 67
  Male | 6 | 6 | 4 | 6 | 4 | 1 | 3 | 3 | 16 | 49

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Outcome Measure: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, Severe TEAEs, Drug-Related TEAEs, and TEAEs Leading to Treatment Discontinuation (Parts 1 and 2 Combined)
Description: An adverse event (AE) was any untoward medical event in a participant who received study drug whether or not the event is considered drug related. TEAEs defined as an AE beginning after first dose of study drug until 28 days after last dose of study drug or existing AEs that worsened after first dose of study drug until the participant's last study visit. Severe AEs defined as incapacitating, inability to perform usual activities. Drug-related TEAEs defined as TEAEs with possible, probable, or definite relationship to study drug. Serious AE criteria included death, life-threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed here. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 16 (End of Study (EoS])
Population: Part 1 and Part 2 Safety Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat 0.7 mg/kg BIW | Roxadustat 0.7 mg/kg TIW | Roxadustat 1.0 mg/kg BIW | Roxadustat 1.0 mg/kg TIW | Roxadustat 1.5 mg/kg BIW | Roxadustat 1.5 mg/kg TIW | Roxadustat 2.0 mg/kg BIW | Roxadustat 2.0 mg/kg TIW | Placebo
Number analyzed (Participants) | 10 | 13 | 12 | 9 | 10 | 11 | 11 | 12 | 28
Participants
  Any TEAEs | 3 | 9 | 7 | 5 | 9 | 7 | 7 | 5 | 13
  Serious TEAEs | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Severe TEAEs | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 1
  Drug-Related TEAEs | 1 | 2 | 2 | 1 | 3 | 3 | 3 | 1 | 3
  TEAEs Leading to Treatment Discontinuation | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1

2. Primary Outcome: Co-Primary Efficacy Outcome Measure: Change From Baseline in Hb at Day 26-29 (End of Treatment)
Description: Mean Hb change from baseline was analyzed by treatment group and study visit. Baseline was defined as the mean of last 3 available values prior to the first dose.
Time Frame: Baseline, End of Treatment (EoT) (Day 26 for TIW Dosing or Day 29 for BIW Dosing)
Population: Part 1 and Part 2 EE Population: Participants who were anemic at baseline (Hb ≤11.0 g/dL and were in study treatment for at least 2.5 weeks with corresponding Hb values. Last-observation-carried-forward (LOCF) method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat 0.7 mg/kg BIW | Roxadustat 0.7 mg/kg TIW | Roxadustat 1.0 mg/kg BIW | Roxadustat 1.0 mg/kg TIW | Roxadustat 1.5 mg/kg BIW | Roxadustat 1.5 mg/kg TIW | Roxadustat 2.0 mg/kg BIW | Roxadustat 2.0 mg/kg TIW | Placebo
Number analyzed (Participants) | 10 | 12 | 5 | 5 | 10 | 11 | 9 | 11 | 23
g/dL
  Baseline | 10.32 (0.678) | 10.03 (0.709) | 9.18 (0.600) | 10.35 (0.849) | 10.28 (0.551) | 10.08 (0.650) | 9.97 (0.430) | 9.93 (0.806) | 10.10 (0.616)
  Change at Day 26-29 | 0.25 (0.849) | 0.60 (0.756) | 0.44 (0.781) | 0.21 (1.016) | 1.22 (1.112) | 1.65 (1.033) | 1.35 (0.577) | 1.75 (1.200) | -0.05 (0.500)
Statistical Analysis 1: Comparison: Roxadustat 0.7 mg/kg BIW vs Placebo; P-value is from inter-group 2-sample t-tests comparing roxadustat change from baseline with placebo change from baseline; Test type: Other; p = 0.2073, t-test, 2 sided — Threshold for significance at 0.05 level
Statistical Analysis 2: Comparison: Roxadustat 0.7 mg/kg TIW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.0046, t-test, 2 sided — Threshold for significance at 0.05 level
Statistical Analysis 3: Comparison: Roxadustat 1.0 mg/kg BIW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.0860, t-test, 2 sided — Threshold for significance at 0.05 level
Statistical Analysis 4: Comparison: Roxadustat 1.0 mg/kg TIW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.4005, t-test, 2 sided — Threshold for significance at 0.05 level
Statistical Analysis 5: Comparison: Roxadustat 1.5 mg/kg BIW vs Placebo; P-value is presented for Day 26-29 timepoint. P-value is from inter-group 2-sample t-tests comparing roxadustat change from baseline with placebo change from baseline; Test type: Other; p < 0.0001, t-test, 2 sided — Threshold for significance at 0.05 level
Statistical Analysis 6: Comparison: Roxadustat 1.5 mg/kg TIW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — Threshold for significance at 0.05 level
Statistical Analysis 7: Comparison: Roxadustat 2.0 mg/kg BIW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — Threshold for significance at 0.05 level
Statistical Analysis 8: Comparison: Roxadustat 2.0 mg/kg TIW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided; Threshold for significance at 0.05 level

3. Primary Outcome: Co-Primary Efficacy Outcome Measure: Change From Baseline in Hb at Week 8 (2 Weeks of Follow Up)
Description: Mean Hb change from baseline was analyzed by treatment group and study visit. Baseline is defined as the mean of last 3 available values prior to the first dose.
Time Frame: Baseline, Week 8 (2 Weeks of Follow Up)
Population: Part 1 and Part 2 EE Population: Participants who were anemic at baseline (Hb ≤11.0 g/dL and were in study treatment for at least 2.5 weeks with corresponding Hb values. LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat 0.7 mg/kg BIW | Roxadustat 0.7 mg/kg TIW | Roxadustat 1.0 mg/kg BIW | Roxadustat 1.0 mg/kg TIW | Roxadustat 1.5 mg/kg BIW | Roxadustat 1.5 mg/kg TIW | Roxadustat 2.0 mg/kg BIW | Roxadustat 2.0 mg/kg TIW | Placebo
Number analyzed (Participants) | 10 | 12 | 5 | 5 | 10 | 11 | 9 | 11 | 23
g/dL
  Baseline | 10.32 (0.678) | 10.03 (0.709) | 9.18 (0.600) | 10.35 (0.849) | 10.28 (0.551) | 10.08 (0.650) | 9.97 (0.430) | 9.93 (0.806) | 10.10 (0.616)
  Change at Week 8 | 0.59 (0.808) | 0.24 (0.846) | 0.50 (0.356) | 0.05 (1.435) | 0.79 (0.916) | 1.31 (0.743) | 1.21 (0.656) | 1.52 (0.815) | 0.04 (0.684)
Statistical Analysis 1: Comparison: Roxadustat 0.7 mg/kg BIW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.0507, t-test, 2 sided — Threshold for significance at 0.05 level
Statistical Analysis 2: Comparison: Roxadustat 0.7 mg/kg TIW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.4502, t-test, 2 sided — Threshold for significance at 0.05 level
Statistical Analysis 3: Comparison: Roxadustat 1.0 mg/kg BIW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other — Threshold for significance at 0.05 level; p = 0.1603, t-test, 2 sided
Statistical Analysis 4: Comparison: Roxadustat 1.0 mg/kg TIW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.9816, t-test, 2 sided — Threshold for significance at 0.05 level
Statistical Analysis 5: Comparison: Roxadustat 1.5 mg/kg BIW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.0139, t-test, 2 sided — Threshold for significance at 0.05 level
Statistical Analysis 6: Comparison: Roxadustat 1.5 mg/kg TIW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — Threshold for significance at 0.05 level
Statistical Analysis 7: Comparison: Roxadustat 2.0 mg/kg BIW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.0001, t-test, 2 sided — Threshold for significance at 0.05 level
Statistical Analysis 8: Comparison: Roxadustat 2.0 mg/kg TIW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — Threshold for significance at 0.05 level

4. Secondary Outcome: Number of Participants With a Hemoglobin Response (Not Due to a RBC Transfusion or IV Iron Supplementation During Treatment)
Description: Hb response defined as an increase in Hb from baseline by ≥1.0 g/dL (not due to red blood cell transfusion or IV iron supplementation during treatment). The baseline for Hb was defined as the mean of the last 3 available Hb values obtained prior to the first dose.
Time Frame: Baseline up to Day 26-29 (EoT), up to Week 8 (2 weeks of follow up), and up to Week 16 (EoS, 4 weeks of follow up)
Population: Part 1 and Part 2 EE Population: Participants who were anemic at baseline (Hb ≤11.0 g/dL) and were in study treatment for at least 2.5 weeks with corresponding Hb values.
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat 0.7 mg/kg BIW | Roxadustat 0.7 mg/kg TIW | Roxadustat 1.0 mg/kg BIW | Roxadustat 1.0 mg/kg TIW | Roxadustat 1.5 mg/kg BIW | Roxadustat 1.5 mg/kg TIW | Roxadustat 2.0 mg/kg BIW | Roxadustat 2.0 mg/kg TIW | Placebo
Number analyzed (Participants) | 10 | 12 | 5 | 5 | 10 | 11 | 9 | 11 | 23
Participants
  Day 26-29 | 1 | 6 | 1 | 1 | 8 | 10 | 7 | 9 | 3
  Week 8 | 5 | 7 | 3 | 2 | 8 | 10 | 9 | 11 | 6
  Week 16 | 7 | 7 | 3 | 2 | 9 | 10 | 9 | 11 | 8

5. Secondary Outcome: Plasma Roxadustat Concentration (Part 2)
Time Frame: Predose on Days 3 (TIW dose groups) or 4 (BIW dose groups), 8, 15, 22, and 26 (TIW dose groups) or 29 (BIW dose groups)
Population: Part 2 PK Population: Participants who received roxadustat and had sufficient plasma data to allow calculation of PK parameters. Participants in the roxadustat groups were evaluated. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable at the specified timepoint.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/milliliter (mL)
Arm/Group | Roxadustat 0.7 mg/kg BIW | Roxadustat 0.7 mg/kg TIW | Roxadustat 1.5 mg/kg BIW | Roxadustat 1.5 mg/kg TIW | Roxadustat 2.0 mg/kg BIW | Roxadustat 2.0 mg/kg TIW
Number analyzed (Participants) | 10 | 13 | 10 | 11 | 9 | 10
nanograms (ng)/milliliter (mL)
  Day 3: number analyzed (Participants) | 0 | 11 | 0 | 11 | 0 | 10
  Day 3 |  | 394.800 (723.156) |  | 260.027 (133.524) |  | 422.700 (148.529)
  Day 4: number analyzed (Participants) | 7 | 0 | 10 | 0 | 9 | 0
  Day 4 | 28.596 (19.737) |  | 168.310 (174.426) |  | 283.067 (376.601) |
  Day 8: number analyzed (Participants) | 9 | 13 | 10 | 11 | 9 | 10
  Day 8 | 19.884 (18.858) | 203.535 (343.167) | 125.185 (223.124) | 168.955 (147.019) | 291.856 (376.910) | 297.500 (393.134)
  Day 15: number analyzed (Participants) | 10 | 12 | 10 | 11 | 9 | 10
  Day 15 | 22.997 (18.442) | 195.483 (369.794) | 134.116 (269.890) | 247.945 (204.624) | 358.400 (491.898) | 175.570 (144.779)
  Day 22: number analyzed (Participants) | 10 | 12 | 10 | 11 | 9 | 10
  Day 22 | 36.432 (33.587) | 153.903 (173.388) | 147.323 (235.302) | 163.100 (167.695) | 171.833 (138.575) | 239.600 (324.307)
  Day 26: number analyzed (Participants) | 0 | 10 | 0 | 10 | 0 | 10
  Day 26 |  | 331.640 (435.773) |  | 223.140 (140.340) |  | 508.889 (295.228)
  Day 29: number analyzed (Participants) | 9 | 0 | 10 | 0 | 9 | 0
  Day 29 | 14.332 (9.935) |  | 150.599 (233.871) |  | 193.622 (279.533) |

6. Secondary Outcome: Change From Baseline in Plasma Erythropoietin in Part 1 Participants at Day 26 or Day 29
Description: Baseline is defined as the last value obtained prior to the first dose.
Time Frame: Baseline (Day 1), 1, 2, 3, 4, 6, 8, 12, 18, 24, 48, and 72 hours on Day 26 (TIW Dosing) or Day 29 (BIW Dosing)
Population: Part 1 Safety Population: Participants who received at least 1 dose of study drug. Participants with missing erythropoietin values at any timepoint were excluded from analysis. Here, 'Number Analyzed' signifies participants evaluable at the specified timepoint.
Measure: Mean (Standard Deviation); unit: milli-international units (mIU)/mL
Arm/Group | Roxadustat 1.0 mg/kg BIW | Roxadustat 1.0 mg/kg TIW | Roxadustat 2.0 mg/kg BIW | Roxadustat 2.0 mg/kg TIW | Placebo
Number analyzed (Participants) | 5 | 3 | 1 | 2 | 6
milli-international units (mIU)/mL
  Day 1, Baseline | 13.46 (5.69) | 13.30 (6.59) | 9.00 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | 8.50 (3.96) | 13.75 (4.53)
  Change at Day 26, 1 Hour: number analyzed (Participants) | 0 | 2 | 0 | 1 | 3
  Change at Day 26, 1 Hour |  | -1.50 (1.41) |  | 0.00 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | 0.17 (0.21)
  Change at Day 26, 2 Hour: number analyzed (Participants) | 0 | 2 | 0 | 1 | 3
  Change at Day 26, 2 Hour |  | -0.85 (1.91) |  | -0.60 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | 0.67 (1.47)
  Change at Day 26, 3 Hour: number analyzed (Participants) | 0 | 2 | 0 | 1 | 3
  Change at Day 26, 3 Hour |  | -0.95 (1.34) |  | 2.30 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | -1.27 (3.15)
  Change at Day 26, 4 Hour: number analyzed (Participants) | 0 | 2 | 0 | 1 | 2
  Change at Day 26, 4 Hour |  | -0.45 (0.07) |  | 29.70 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | 0.50 (4.24)
  Change at Day 26, 6 Hour: number analyzed (Participants) | 0 | 2 | 0 | 1 | 3
  Change at Day 26, 6 Hour |  | 8.05 (11.81) |  | 132.80 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | 0.33 (3.80)
  Change at Day 26, 8 Hour: number analyzed (Participants) | 0 | 2 | 0 | 1 | 3
  Change at Day 26, 8 Hour |  | 57.95 (63.29) |  | 462.00 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | 0.20 (1.18)
  Change at Day 26, 12 Hour: number analyzed (Participants) | 0 | 2 | 0 | 2 | 3
  Change at Day 26, 12 Hour |  | 81.80 (81.03) |  | 492.00 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | -1.30 (1.71)
  Change at Day 26, 18 Hour: number analyzed (Participants) | 0 | 2 | 0 | 1 | 3
  Change at Day 26, 18 Hour |  | 37.30 (13.01) |  | 176.90 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | 0.87 (1.07)
  Change at Day 26, 24 Hour: number analyzed (Participants) | 0 | 2 | 0 | 1 | 3
  Change at Day 26, 24 Hour |  | 22.35 (19.73) |  | 33.90 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | 2.60 (5.46)
  Change at Day 26, 48 Hour: number analyzed (Participants) | 0 | 2 | 0 | 1 | 2
  Change at Day 26, 48 Hour |  | 0.55 (10.39) |  | -0.50 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | -7.50 (2.40)
  Change at Day 26, 72 Hour: number analyzed (Participants) | 0 | 2 | 0 | 1 | 2
  Change at Day 26, 72 Hour |  | -2.85 (5.02) |  | -1.50 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | -0.60 (1.27)
  Change at Day 29, 1 Hour: number analyzed (Participants) | 4 | 0 | 0 | 0 | 3
  Change at Day 29, 1 Hour | -1.08 (1.22) |  |  |  | -1.57 (1.14)
  Change at Day 29, 2 Hour: number analyzed (Participants) | 4 | 0 | 0 | 0 | 3
  Change at Day 29, 2 Hour | -1.27 (2.23) |  |  |  | -2.73 (1.85)
  Change at Day 29, 3 Hour: number analyzed (Participants) | 4 | 0 | 0 | 0 | 3
  Change at Day 29, 3 Hour | -0.55 (1.13) |  |  |  | -3.70 (2.14)
  Change at Day 29, 4 Hour: number analyzed (Participants) | 4 | 0 | 0 | 0 | 3
  Change at Day 29, 4 Hour | 12.03 (10.12) |  |  |  | -4.90 (1.95)
  Change at Day 29, 6 Hour: number analyzed (Participants) | 4 | 0 | 0 | 0 | 3
  Change at Day 29, 6 Hour | 66.85 (43.07) |  |  |  | -4.17 (1.27)
  Change at Day 29, 8 Hour: number analyzed (Participants) | 4 | 0 | 0 | 0 | 3
  Change at Day 29, 8 Hour | 135.08 (83.95) |  |  |  | -2.97 (2.20)
  Change at Day 29, 12 Hour: number analyzed (Participants) | 4 | 0 | 0 | 0 | 3
  Change at Day 29, 12 Hour | 77.35 (43.80) |  |  |  | -2.07 (1.08)
  Change at Day 29, 18 Hour: number analyzed (Participants) | 4 | 0 | 0 | 0 | 3
  Change at Day 29, 18 Hour | 43.80 (13.41) |  |  |  | -0.20 (1.77)
  Change at Day 29, 24 Hour: number analyzed (Participants) | 4 | 0 | 0 | 0 | 3
  Change at Day 29, 24 Hour | 10.18 (3.16) |  |  |  | -3.07 (0.96)
  Change at Day 29, 48 Hour: number analyzed (Participants) | 3 | 0 | 0 | 0 | 3
  Change at Day 29, 48 Hour | -5.17 (4.70) |  |  |  | -4.87 (2.24)
  Change at Day 29, 72 Hour: number analyzed (Participants) | 4 | 0 | 0 | 0 | 3
  Change at Day 29, 72 Hour | -2.93 (3.91) |  |  |  | -1.63 (4.71)

7. Secondary Outcome: Change From Baseline in Plasma Erythropoietin in Part 2 Participants at 4, 8, 12, and 24 Hours on Day 1
Description: Baseline is defined as the last value obtained prior to the first dose.
Time Frame: Baseline, 4, 8, 12, and 24 hours on Day 1
Population: Part 2 PK Population: Participants who received roxadustat and had sufficient plasma data to allow calculation of PK parameters. Participants with missing erythropoietin values at any timepoint were excluded from analysis.
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Roxadustat 0.7 mg/kg BIW | Roxadustat 0.7 mg/kg TIW | Roxadustat 1.5 mg/kg BIW | Roxadustat 1.5 mg/kg TIW | Roxadustat 2.0 mg/kg BIW | Roxadustat 2.0 mg/kg TIW | Placebo
Number analyzed (Participants) | 0 | 2 | 2 | 0 | 2 | 0 | 0
mIU/mL
  Baseline |  | 8.30 (2.26) | 9.55 (3.32) |  | 10.45 (4.31) |  |
  Change at 4 Hour |  | 2.80 (3.96) | 2.10 (3.54) |  | 1.00 (2.97) |  |
  Change at 8 Hour |  | 66.70 (90.23) | 100.40 (92.77) |  | 42.05 (36.98) |  |
  Change at 12 Hour |  | 66.25 (90.16) | 147.15 (128.91) |  | 201.10 (240.42) |  |
  Change at 24 Hour |  | 10.05 (8.56) | 107.65 (53.25) |  | 461.05 (589.80) |  |

ADVERSE EVENTS:
Time Frame: Baseline up to Week 16 (EoS)
Description: Part 1 and Part 2 Safety Population: Participants who received at least 1 dose of study drug.
Arm/Group | Roxadustat 0.7 mg/kg BIW | Roxadustat 0.7 mg/kg TIW | Roxadustat 1.0 mg/kg BIW | Roxadustat 1.0 mg/kg TIW | Roxadustat 1.5 mg/kg BIW | Roxadustat 1.5 mg/kg TIW | Roxadustat 2.0 mg/kg BIW | Roxadustat 2.0 mg/kg TIW | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 4/13 | 0/12 | 0/9 | 0/10 | 0/11 | 0/11 | 0/12 | 1/28
Other Adverse Events (participants affected / at risk) | 3/10 | 9/13 | 7/12 | 5/9 | 9/10 | 7/11 | 7/11 | 5/12 | 12/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roxadustat 0.7 mg/kg BIW (N=10) | Roxadustat 0.7 mg/kg TIW (N=13) | Roxadustat 1.0 mg/kg BIW (N=12) | Roxadustat 1.0 mg/kg TIW (N=9) | Roxadustat 1.5 mg/kg BIW (N=10) | Roxadustat 1.5 mg/kg TIW (N=11) | Roxadustat 2.0 mg/kg BIW (N=11) | Roxadustat 2.0 mg/kg TIW (N=12) | Placebo (N=28)
Arteriovenous fistula site (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Roxadustat 0.7 mg/kg BIW (N=10) | Roxadustat 0.7 mg/kg TIW (N=13) | Roxadustat 1.0 mg/kg BIW (N=12) | Roxadustat 1.0 mg/kg TIW (N=9) | Roxadustat 1.5 mg/kg BIW (N=10) | Roxadustat 1.5 mg/kg TIW (N=11) | Roxadustat 2.0 mg/kg BIW (N=11) | Roxadustat 2.0 mg/kg TIW (N=12) | Placebo (N=28)
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 2 | 1 | 1 | 0 | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram poor R-wave progression (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram repolarisation abnormality (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0/6 | 0/6 | 0/4 | 1/6 | 0/4 | 0/1 | 0/3 | 0/3 | 0/16 — This is a sex-specific adverse event that only affects male participants.
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gallbladder polyp (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other